CLINICAL TRIAL: NCT02091739
Title: Prospective, Randomized, Double-blind, Placebo-controlled, Parallel-group Multicenter Study, With an Extension Period of Dose-blinded Active Treatment, to Investigate the Efficacy and Safety of Two Dose Levels of NT 201 in Treating Chronic Troublesome Sialorrhea in Various Neurological Conditions
Brief Title: Clinical Study to Investigate the Efficacy and Safety of Two Dose Levels of NT 201 Versus Placebo in Treating Chronic Troublesome Sialorrhea in Various Neurological Conditions
Acronym: SIAXI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ60201_3090_1; 2012-005539-10 (EudraCT Number)
Record Dates: First submitted 2014-03-18; First posted 2014-03-19 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-01

CONDITIONS: Chronic Troublesome Sialorrhea; Parkinson's Disease; Post-stroke; Traumatic Brain Injury
MeSH Terms: conditions — Parkinson Disease; Brain Injuries, Traumatic | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IncobotulinumtoxinA (Xeomin) (100 Units) (Experimental): * Main period (1 treatment cycle): Subjects to receive 100 Units.
  * Extension period (3 treatment cycles): Subjects to receive 100 Units per treatment cycle.
  * Mode of administration: Four injections per treatment cycle (parotid and submandibular glands, bilateral)
  Interventions: Drug: IncobotulinumtoxinA (100 Units)
- IncobotulinumtoxinA (Xeomin) (75 Units) (Experimental): * Main period (1 treatment cycle): Subjects to receive 75 Units.
  * Extension period (3 treatment cycles): Subjects to receive 75 Units per treatment cycle.
  * Mode of administration: Four injections per treatment cycle (parotid and submandibular glands, bilateral)
  Interventions: Drug: IncobotulinumtoxinA (75 Units)
- Placebo (Placebo Comparator): * Main period (1 treatment cycle): Subjects to receive placebo injection.
  * Extension period (3 treatment cycles): Subjects will be randomized to receive either 75 or 100 Units IncobotulinumtoxinA per treatment cycle.
  * Mode of administration: Four injections per treatment cycle (parotid and submandibular glands, bilateral)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IncobotulinumtoxinA (100 Units) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: IncobotulinumtoxinA (Xeomin) (100 Units)
Drug: IncobotulinumtoxinA (75 Units) — Active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins. Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Other Names: Xeomin; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: IncobotulinumtoxinA (Xeomin) (75 Units)
Drug: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the efficacy and safety of two different dose levels of NT 201 (75 U or 100 U per cycle), compared with placebo, in reducing the salivary flow rate, and the severity and frequency of chronic troublesome sialorrhea that occurs as a result of various neurological conditions in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of the basic neurological condition associated with sialorrhea (as above, (i), (ii) or (iii); with onset at least 6 months before screening).
* Chronic troublesome sialorrhea related to parkinsonism or stroke or traumatic brain injury (for at least 3 months) at screening, defined as the presence of all of the following, at screening and at baseline and for at least the 3 months before screening (where retrospective response to questionnaires is impossible, a statement of equivalent severity will suffice):

  1. A Drooling Severity and Frequency Scale [DSFS] sum score of at least 6 points and
  2. A score of at least 2 points for each item of the DSFS and
  3. A score of at least 3 points on the modified Radboud Oral Motor Inventory for Parkinson's Disease [mROMP], Section 'III Drooling', Item A).
* A score of at most 2 points on the mROMP Section 'II Swallowing Symptoms' Item A) and a score of at most 3 points on Item C), at screening and at baseline.

Exclusion Criteria:

* Non-neurological secondary causes of sialorrhea.
* Unstable concomitant medication influencing sialorrhea (such as anticholinergics for the treatment of parkinsonism; dosages of these medications must have been stable for at least 4 weeks before study entry, i.e. screening, and must be planned to remain stable during the course of the study.
* Recent (i.e., four weeks) drug treatment for sialorrhea.
* History of recurrent aspiration pneumonia.
* Extremely poor dental/oral condition as assessed by a qualified dentist.
* Recent (i.e., one year for sialorrhea, 14 weeks for other indications) treatment with - or known hypersensitivity to - Botulinum toxin, or known hypersensitivity to any ingredient of the study preparation.
* Recent (i.e., four weeks) changes in anti-parkinsonian medication.
* Previous or planned surgery or irradiation to control sialorrhea.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (31):
- Germany (11):
  - Merz investigational site #049172, Bonn
  - Merz Investigational Site #049335, Gera
  - Merz Investigational Site #049337, Haag i.OB
  - Merz Investigational Site #049072, Munich
  - Merz Investigational Site #049148, Munich
  - Merz Investigational Site #049300, Nümbrecht
  - Merz Investigational Site #049303, Regensburg
  - Merz investigational site #049348, Stadtroda
  - Merz Investigational Site #049143, Ulm
  - Merz Investigational Site #049333, Wolfach
  - Merz Investigational Site #049302, Würzburg
- Poland (20):
  - Merz investigational site #048068, Bydgoszcz
  - Merz Investigational Site #048088, Bydgoszcz
  - Merz Investigational Site #048029, Gdansk
  - Merz investigational site #048074, Gdansk
  - Merz investigational site #048078, Jaworzno
  - Merz investigational site #048076, Katowice
  - Merz investigational site #048077, Katowice
  - Merz investigational Site #048067, Kielce
  - Merz investigational site #048059, Krakow
  - Merz investigational site #048031, Krakow
  - Merz Investigational Site #048087, Krakow
  - Merz Investigational Site #048022, Lodz
  - Merz investigational site #048070, Lublin
  - Merz investigational site #048085, Lublin
  - Merz investigational site #048072, Luboń
  - Merz Investigational Site #048075, Sandomierz
  - Merz Investigational Site #048086, Torun
  - Merz investigational site #048065, Warsaw
  - Merz investigational site #048056, Warsaw
  - Merz investigational site #048064, Warsaw

REFERENCES:
- [Derived] Jost WH, Friedman A, Michel O, Oehlwein C, Slawek J, Bogucki A, Ochudlo S, Banach M, Pagan F, Flatau-Baque B, Dorsch U, Csikos J, Blitzer A. Long-term incobotulinumtoxinA treatment for chronic sialorrhea: Efficacy and safety over 64 weeks. Parkinsonism Relat Disord. 2020 Jan;70:23-30. doi: 10.1016/j.parkreldis.2019.11.024. Epub 2019 Nov 26. PMID 31794936
- [Derived] Jost WH, Friedman A, Michel O, Oehlwein C, Slawek J, Bogucki A, Ochudlo S, Banach M, Pagan F, Flatau-Baque B, Csikos J, Cairney CJ, Blitzer A. SIAXI: Placebo-controlled, randomized, double-blind study of incobotulinumtoxinA for sialorrhea. Neurology. 2019 Apr 23;92(17):e1982-e1991. doi: 10.1212/WNL.0000000000007368. Epub 2019 Mar 27. PMID 30918101

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 12 sites in Poland and Germany.
Pre-assignment Details: A total of 216 participants were screened for the study, of which 184 participants were randomized and treated in the Main Period (MP) of the study. A total of 173 participants who completed the MP, entered the 2 treatment arms of the Extension Period (EP) of the study.
Groups:
- Placebo: Participants received one injection session of overall 2.0 milliliter (mL) placebo matched to the volume of incobotulinumtoxinA via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 in the MP.
- MP: IncobotulinumtoxinA (Xeomin) (75 Units): Participants received one injection session of overall 2.0 mL incobotulinumtoxinA containing 75 units via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 in the MP.
- MP: IncobotulinumtoxinA (Xeomin) (100 Units): Participants received one injection session of overall 2.0 mL incobotulinumtoxinA containing 100 units via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 in the MP.
- EP: IncobotulinumtoxinA (Xeomin) (75 Units): Participants received overall 2.0 mL incobotulinumtoxinA containing 75 units via bilateral intraglandular injection into the parotid and submandibular glands at each of the three injection sessions in the EP.
- EP: IncobotulinumtoxinA (Xeomin) (100 Units): Participants received overall 2.0 mL incobotulinumtoxinA containing 100 units via bilateral intraglandular injection into the parotid and submandibular glands at each of the three injection sessions in the EP.
Period: MP: 16 Weeks
Arm/Group | Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units) | EP: IncobotulinumtoxinA (Xeomin) (75 Units) | EP: IncobotulinumtoxinA (Xeomin) (100 Units)
Started | 36 | 74 | 74 | 0 | 0
Completed | 32 | 69 | 72 | 0 | 0
Not Completed | 4 | 5 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Period: EP: 48 Weeks
Arm/Group | Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units) | EP: IncobotulinumtoxinA (Xeomin) (75 Units) | EP: IncobotulinumtoxinA (Xeomin) (100 Units)
Started | 0 | 0 | 0 | 84 | 89
Completed (Participants who completed the MP (n=173), entered the 2 treatment arms of the EP of the study.) | 0 | 0 | 0 | 76 | 75
Not Completed | 0 | 0 | 0 | 8 | 14
Not completed — Other | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) is the subset of participants who were treated and had at least the baseline value of unstimulated salivary flow (uSFR).
Groups:
- MP: Placebo: Participants received one injection session of overall 2.0 mL placebo matched to the volume of incobotulinumtoxinA via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 in the MP.
- Total: Total of all reporting groups
Arm/Group | MP: Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units) | Total
Number analyzed (Participants) | 36 | 74 | 74 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 30 | 28 | 77
  >=65 years | 17 | 44 | 46 | 107
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 24 | 22 | 54
  Male | 28 | 50 | 52 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 36 | 74 | 73 | 183
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 36 | 74 | 73 | 183
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 80.6 (16.4) | 78.4 (17.1) | 79.8 (14) | 79.4 (15.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 28.5 (6) | 26.7 (5.2) | 27.7 (3.8) | 27.5 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: MP: Change From Baseline in Unstimulated Salivary Flow (uSFR) Rate at Week 4
Description: uSFR was assessed by weighing of dental rolls soaked with saliva over 5 minutes and then procedure was repeated after 30 minutes and the average of the 2 results for flow rate was calculated.
Time Frame: Baseline and Week 4
Population: Analysis covers all participants from FAS who have at least one post-baseline uSFR assessment. The FAS is the subset of participants who were treated and had at least the baseline value of uSFR.
Measure: Least Squares Mean (Standard Error); unit: gram per minute (g/min)
Arm/Group | MP: Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units)
Number analyzed (Participants) | 36 | 73 | 73
gram per minute (g/min) | -0.04 (0.033) | -0.06 (0.027) | -0.13 (0.026)
Statistical Analysis 1: Comparison: MP: Placebo vs MP: IncobotulinumtoxinA (Xeomin) (100 Units); A fixed sequence test procedure was used for the confirmatory analysis of the co-primary endpoints by comparing the least square (LS) means estimates of an mixed model repeated measurement (MMRM) model (2-sided, significance level alpha=0.05) between treatment groups in the following order: 1. IncobotulinumtoxinA 100 units versus (v) Placebo 2. IncobotulinumtoxinA 75 units v Placebo; Test type: Superiority; p = 0.004, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.15 to 0.03], Standard Error of Mean 0.031
Statistical Analysis 2: Comparison: MP: Placebo vs MP: IncobotulinumtoxinA (Xeomin) (75 Units); A fixed sequence test procedure was used for the confirmatory analysis of the co-primary endpoints by comparing the least square means estimates of an MMRM model (2-sided, significance level alpha=0.05) between treatment groups in the following order: 1. IncobotulinumtoxinA 100 units v Placebo 2. IncobotulinumtoxinA 75 units v Placebo; Test type: Superiority; p = 0.542, MMRM; LS mean difference = -0.02, 95% CI 2-sided [-0.08 to 0.04], Standard Error of Mean 0.03

2. Primary Outcome: MP: Participant's Global Impression of Change Scale (GICS) at Week 4
Description: The GICS was used to measure the impression of change due to treatment. The response option was a common 7-point Likert scale that ranged from -3 = very much worse to +3 = very much improved and was applicable for participant and caregiver. If the participant was not able to answer then carer's rating was to be recorded instead of participant's rating and the participant's rating was left blank.
Time Frame: Week 4
Population: The FAS is the subset of participants who were treated and had at least the baseline value of uSFR.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MP: Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units)
Number analyzed (Participants) | 36 | 74 | 74
units on a scale | 0.67 (0.186) | 1.02 (0.148) | 1.25 (0.144)
Statistical Analysis 1: Comparison: MP: Placebo vs MP: IncobotulinumtoxinA (Xeomin) (100 Units); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.002, MMRM; LS mean difference = 0.58, 95% CI 2-sided [0.22 to 0.94], Standard Error of Mean 0.183
Statistical Analysis 2: Comparison: MP: Placebo vs MP: IncobotulinumtoxinA (Xeomin) (75 Units); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.055, MMRM; LS mean difference = 0.35, 95% CI 2-sided [-0.01 to 0.71], Standard Error of Mean 0.181

3. Secondary Outcome: MP: Change From Baseline in Unstimulated Salivary Flow (uSFR) Rate at Week 8 and 12
Description: as for outcome 1
Time Frame: Baseline, Week 8 and 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: g/min
Arm/Group | MP: Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units)
Number analyzed (Participants) | 36 | 73 | 73
g/min
  Week 8 | -0.02 (0.033) | -0.08 (0.027) | -0.13 (0.026)
  Week 12 | -0.03 (0.033) | -0.1 (0.027) | -0.12 (0.026)

4. Secondary Outcome: MP: Global Impression of Change Scale (GICS) at Week 1, 2, 8 and 12
Description: The GICS was used to measure the investigator's impression of change due to treatment. The response option was a common 7-point Likert scale that ranged from -3 = very much worse to +3 = very much improved and was applicable for participant and caregiver. If the participant was not able to answer then carer's rating was to be recorded instead of participant's rating and the participant's rating was left blank.
Time Frame: Week 1, 2, 8, and 12
Population: The FAS is the subset of participants who were treated and had at least the baseline value of uSFR.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | MP: Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units)
Number analyzed (Participants) | 36 | 74 | 74
units on a scale
  Week 1 | 0.67 (0.17) | 0.73 (0.138) | 0.96 (0.133)
  Week 2 | 0.83 (0.178) | 0.91 (0.143) | 1.11 (0.139)
  Week 8 | 0.47 (0.192) | 1.07 (0.151) | 1.3 (0.148)
  Week 12 | 0.56 (0.197) | 0.98 (0.156) | 1.21 (0.152)

ADVERSE EVENTS:
Time Frame: MP: From first injection up to first injection in EP (Week 16). EP: From first injection in EP (Week 16) up to end of study (Week 64).
Description: The investigator asked the participant for adverse events systematically at each visit. Two participants received the wrong or no dose in single EP cycles due to procedural reasons and hence were not included in the safety analyses that cover the complete EP: IncobotulinumtoxinA (Xeomin) (75 Units) arm.
Groups:
- Placebo: Participants received one injection session of overall 2.0 mL placebo matched to the volume of incobotulinumtoxinA via bilateral intraglandular injection into the parotid and submandibular glands on Day 1 in the MP.
Arm/Group | Placebo | MP: IncobotulinumtoxinA (Xeomin) (75 Units) | MP: IncobotulinumtoxinA (Xeomin) (100 Units) | EP: IncobotulinumtoxinA (Xeomin) (75 Units) | EP: IncobotulinumtoxinA (Xeomin) (100 Units)
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/74 | 0/74 | 3/82 | 2/89
Serious Adverse Events (participants affected / at risk) | 3/36 | 6/74 | 9/74 | 15/82 | 14/89
Other Adverse Events (participants affected / at risk) | 2/36 | 14/74 | 10/74 | 22/82 | 22/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | MP: IncobotulinumtoxinA (Xeomin) (75 Units) (N=74) | MP: IncobotulinumtoxinA (Xeomin) (100 Units) (N=74) | EP: IncobotulinumtoxinA (Xeomin) (75 Units) (N=82) | EP: IncobotulinumtoxinA (Xeomin) (100 Units) (N=89)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device battery replacement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medical device change (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angioplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterostomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Explorative laparotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laparotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal stone removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureter dilation procedure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dopamine dysregulation syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angiogram (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (8) | 2 (2)
Drop attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Freezing phenomenon (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Akinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac pacemaker insertion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Faecal vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Giant cell epulis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Extravasation of urine (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=36) | MP: IncobotulinumtoxinA (Xeomin) (75 Units) (N=74) | MP: IncobotulinumtoxinA (Xeomin) (100 Units) (N=74) | EP: IncobotulinumtoxinA (Xeomin) (75 Units) (N=82) | EP: IncobotulinumtoxinA (Xeomin) (100 Units) (N=89)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 6 (8) | 2 (5) | 5 (9) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 4 (5) | 0 (0) | 3 (3) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 4 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 4 (5) | 3 (3) | 3 (4) | 10 (13)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.